CLINICAL TRIAL: NCT01915095
Title: Enhancement of Hand Motor Function After Cervical Spinal Cord Injury
Brief Title: Improving Motor Function After Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: B0815-R; NCT02701790 (obsolete NCT alias)
Record Dates: First submitted 2013-07-19; First posted 2013-08-02 (Estimated); Results first posted 2020-11-04 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; neural control; motor function; hand movement
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Motor task+ Magnetic stimulation (Active Comparator): Participants will be asked to complete a precision grip with the index and thumb finger at the same time as flexing or extending the wrist. magnetic stimulation to the brain will be administered and measurements will be taken during movement.
  Interventions: Device: rTMS; Device: Sham rTMS; Other: Motor Task
- rTMS/sham rTMS (Active Comparator): Participant will be randomly assigned to one of 3 groups: repetitive transcranial magnetic stimulation (rTMS), sham (fake) rTMS, or sham (fake) rTMS over control brain area will be administered to the brain. the stimulation will be targeting finger and wrist muscles during movement.
  Interventions: Device: rTMS; Device: Sham rTMS
- Training + rTMS/ Sham rTMS (Active Comparator): Participants will be asked to follow a target line on the computer as accurately as possible while performing precision grips or foot movement . Magnetic stimulation will be given during rest and movement.
  Interventions: Device: rTMS; Device: Sham rTMS; Other: Training

INTERVENTIONS:
Device: rTMS — small magnetic pulses will be given to the brain in a non invasive manner.
Device: Sham rTMS — sham or fake stimulation (TMS or rTMS) will be given to the brain in a non invasive manner
Other: Training — at the direction of the researcher the participant will be instructed to do repetitive motor movements with their arm, hand or leg. this is called training
  Arms: Training + rTMS/ Sham rTMS
Other: Motor Task — participants will be asked to perform specific motor tasks or movements with their fingers, hands, arms or legs.
  Arms: Motor task+ Magnetic stimulation

SUMMARY:
The goals of this study are to examine the physiology of Central Nervous System pathways contributing to the control of upper and lower extremity movements after SCI, and to promote the recovery of extremity movements by using non-invasive brain stimulation and motor training.

DETAILED DESCRIPTION:
This study will consist of electromyography (surface and intramuscular), peripheral nerve stimulation, and transcranial magnetic stimulation, electrical stimulation, of the hand, arm, leg, and foot representation of the primary motor cortex, as well as MRI scans of the brain. The investigators will examine the physiological measurements of upper and lower extremity muscles (such as in the first dorsal interosseous (FDI), biceps brachii (BIC), anterior deltoid (AD), tibialis anterior (TA), hamstring (HAMS) and quadriceps (QUAD)). This study may occur at the Miami Project to cure Paralysis at the University of Miami. The investigators will include subjects between the ages of 18 and 85, both healthy controls and individuals with chronic spinal cord injuries that occurred at least 6 months prior to recruitment. Both healthy controls and those with spinal cord injuries will be able to perform small hand and arm movements and small leg and foot movements. The primary outcome measures of this study are muscle responses to stimulation with magnetic pulses using TMS and electrical stimulation of a peripheral nerve in the arm or leg. The investigators propose to enhance the recovery of motor function by using new protocols of high frequency non-invasive repetitive TMS (rTMS) and motor training. Repetitive TMS will be used during hand, arm, leg and foot movements in a task-dependent manner to induce cortical plasticity and enhance voluntary output of the muscles associated with those movements. Second, rTMS will be applied in a task-dependent manner during a visuo-motor training task that also involves movements of the hands, arms, legs or feet.

ELIGIBILITY:
Inclusion Criteria:

Male and female Veterans and non Veterans with spinal cord injury at least 6 months after injury was sustained. The investigators also plan to enroll control subjects who do not have any history of spinal cord injury.

Participants who are unimpaired healthy controls:

* Male and females between ages 18-85 years
* Right handed
* Able to complete precision grips with both hands
* Able to complete full wrist flexion-extension bilaterally
* Able to walk unassisted
* Able to complete full ankle flexion-extension bilaterally

Participants who have had a spinal cord injury:

* Male and females between ages 18-85 years
* Chronic SCI ( 6 months of injury)
* Spinal Cord injury at or above L5
* The ability to produce a visible precision grip force with one hand
* Individuals who have the ability to pick up a small object (large paperclip) from a table independently
* Able to perform some small wrist flexion and extension (measured by a goniometer)
* The ability to perform a small visible contraction with dorsiflexor and hip flexor muscles
* No subjects will be excluded based on their race, religion, ethnicity, gender or HIV status.

Exclusion Criteria:

Exclusion criteria for enrollment For SCI and Healthy Control Subjects (for stimulation):

* Uncontrolled medical problems including pulmonary, cardiovascular or orthopedic disease
* Any debilitating disease prior to the SCI that caused exercise intolerance
* Premorbid, ongoing major depression or psychosis, altered cognitive status
* History of head injury or stroke
* Metal plate in skull
* History of seizures
* Receiving drugs acting primarily on the central nervous system, which lower the seizure threshold (see appendix 2)
* Pregnant females
* Ongoing cord compression or a syrinx in the spinal cord or who suffer from a spinal cord disease such as spinal stenosis, spina bifida, MS, or herniated cervical disk
* Individuals with scalp shrapnel, cochlear implants, or aneurysm clips.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica A Perez, PhD, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (3):
- United States (3):
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Wrist Flexion and Precision Grip + rTMS and Sham rTMS: This study arm is a crossover design. Participants will complete the following two randomized sessions: 1. Wrist flexion and precision grip + rTMS; 2. Wrist flexion and precision grip + Sham rTMS.
  Participants will complete two study visits each lasting ~2 hours separated by at least two days.
  In the Wrist flexion and precision grip + rTMS study visit, participants are asked to complete a precision grip with the index and thumb finger at the same time as flexing the wrist. Transcranial magnetic stimuli (TMS) to the brain will be administered and TMS measurements in the form of motor evoked potentials (MEPs) will be taken at minute 0, 10, 30, and 60.
  Wrist flexion and precision grip + Sham rTMS:
  The same procedures listed above will be completed before and after Sham rTMS.
- Wrist Extension and Precision Grip + rTMS and Sham rTMS: This study arm is a crossover design. Participants will complete the following two randomized sessions: 1. Wrist extension and precision grip + rTMS; 2. Wrist extension and precision grip + Sham rTMS.
  Participants will complete two study visits each lasting ~2 hours separated by at least two days.
  In the Wrist extension and precision grip + rTMS study visit, participants are asked to complete a precision grip with the index and thumb finger at the same time as extending the wrist. Transcranial magnetic stimuli (TMS) to the brain will be administered and TMS measurements in the form of motor evoked potentials (MEPs) will be taken at minute 0, 10, 30, and 60.
  Wrist extension and precision grip + Sham rTMS:
  The same procedures listed above will be completed before and after Sham rTMS.
- rTMS/Sham rTMS/Sham rTMS Over Control Brain Area: This study arm is a 3 way crossover design. Participants are randomized to one of the 3 study groups: rTMS, Sham rTMS, and Sham rTMS over control brain area. Participants will complete all study groups. Each study group consists of one study visit lasting ~2 hours and there is a 1 week washout period between each study visit.
  rTMS stimulation: In this group, rTMS stimulation will be targeting finger and wrist muscles during precision grip. TMS measurements in the form of motor evoked potentials (MEPs) will be taken at minute 0, 10, 30, and 60. The maximum voluntary contraction (MVC) will be measured using surface EMG before rTMS and again after.
  Sham or fake rTMS stimulation: In this group, Sham rTMS stimulation will be targeting finger and wrist muscles during precision grip. TMS measurements in the form of MEPs will be taken at minute 0, 10, 30, and 60. The MVC will be measured using surface EMG before rTMS and again after.
  Sham rTMS over control brain area: In this group, Sham rTMS will be applies over the dorsolateral prefrontal cortex (DLPFC) or at the leg presentation of the primary motor cortex, or at other related control area. TMS measurements in the form of MEPs will be taken at minute 0, 10, 30, and 60. The MVC will be measured using surface EMG before rTMS and again after.
  Participants are asked to wait a 1 week washout period between sessions.
- Training + rTMS: Participants are asked to follow a target line on the computer as accurately as possible while performing precision grips. Magnetic stimulation will be given during. Participants are asked to complete 10 of these sessions. Participants will also be asked to complete measurements at Baseline, Post 5 sessions, and Post all training sessions.
- Training + Sham rTMS: Participants are asked to follow a target line on the computer as accurately as possible while performing precision grips. Sham or fake Magnetic stimulation will be given during. Participants are asked to complete 10 of these sessions. Participants will also be asked to complete measurements at Baseline, Post 5 sessions, and Post all training sessions.
Period: Overall Study
Arm/Group | Wrist Flexion and Precision Grip + rTMS and Sham rTMS | Wrist Extension and Precision Grip + rTMS and Sham rTMS | rTMS/Sham rTMS/Sham rTMS Over Control Brain Area | Training + rTMS | Training + Sham rTMS
Started | 10 | 10 | 5 | 8 | 9
SCI | 5 | 5 | 5 | 8 | 9
Control | 5 | 5 | 0 | 0 | 0
Completed | 10 | 10 | 5 | 4 | 3
Not Completed | 0 | 0 | 0 | 4 | 6
Not completed — Some subjects were unable to commit to the training study. | 0 | 0 | 0 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Wrist Flexion and Precision Grip + rTMS and Sham rTMS (SCI); Wrist Flexion and Precision Grip + rTMS and Sham rTMS (Controls): This study arm is a crossover design. Participants will complete the following two randomized sessions: 1. Wrist flexion and precision grip + rTMS; 2. Wrist flexion and precision grip + Sham rTMS.
  Participants will complete two study visits each lasting ~2 hours separated by at least two days.
  In the Wrist flexion and precision grip + rTMS study visit, participants are asked to complete a precision grip with the index and thumb finger at the same time as flexing the wrist. Transcranial magnetic stimuli (TMS) to the brain will be administered and TMS measurements in the form of motor evoked potentials (MEPs) will be taken at minute 0, 10, 30, and 60.
  Wrist flexion and precision grip + Sham rTMS:
  The same procedures listed above will be completed before and after Sham rTMS.
- Wrist Extension and Precision Grip + rTMS and Sham rTMS (SCI); Wrist Extension and Precision Grip + rTMS and Sham rTMS (Controls): This study arm is a crossover design. Participants will complete the following two randomized sessions: 1. Wrist extension and precision grip + rTMS; 2. Wrist extension and precision grip + Sham rTMS.
  Participants will complete two study visits each lasting ~2 hours separated by at least two days.
  In the Wrist extension and precision grip + rTMS study visit, participants are asked to complete a precision grip with the index and thumb finger at the same time as extending the wrist. Transcranial magnetic stimuli (TMS) to the brain will be administered and TMS measurements in the form of motor evoked potentials (MEPs) will be taken at minute 0, 10, 30, and 60.
  Wrist extension and precision grip + Sham rTMS:
  The same procedures listed above will be completed before and after Sham rTMS.
- Training + rTMS: Participants will be asked to follow a target line on the computer as accurately as possible while performing precision grips or foot movement . Magnetic stimulation will be given during rest and movement.
  rTMS: small magnetic pulses will be given to the brain in a non invasive manner.
  Training: at the direction of the researcher the participant will be instructed to do repetitive motor movements with their arm, hand or leg. this is called training
- Training + Sham rTMS: Participants will be asked to follow a target line on the computer as accurately as possible while performing precision grips or foot movement . Magnetic stimulation will be given during rest and movement.
  Sham rTMS: sham or fake stimulation (TMS or rTMS) will be given to the brain in a non invasive manner
  Training: at the direction of the researcher the participant will be instructed to do repetitive motor movements with their arm, hand or leg. this is called training
- Total: Total of all reporting groups
Arm/Group | Wrist Flexion and Precision Grip + rTMS and Sham rTMS (SCI) | Wrist Flexion and Precision Grip + rTMS and Sham rTMS (Controls) | Wrist Extension and Precision Grip + rTMS and Sham rTMS (SCI) | Wrist Extension and Precision Grip + rTMS and Sham rTMS (Controls) | rTMS/Sham rTMS/Sham rTMS Over Control Brain Area | Training + rTMS | Training + Sham rTMS | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 4 | 3 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 5 | 5 | 5 | 4 | 3 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 44 [30 to 58] | 48 [26 to 56] | 53 [37 to 58] | 51 [41 to 56] | 43 [23 to 61] | 45 [33 to 56] | 41 [30 to 55] | 45 [23 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 3 | 1 | 1 | 1 | 0 | 8
  Male | 5 | 3 | 2 | 4 | 4 | 3 | 3 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 4 | 1 | 4 | 3 | 2 | 21
  Not Hispanic or Latino | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 8
  Unknown or Not Reported | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Black or African American | 1 | 3 | 1 | 2 | 3 | 2 | 2 | 14
  White | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 4
  More than one race | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 8
  Unknown or Not Reported | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 5 | 5 | 5 | 4 | 3 | 32

OUTCOME MEASURES:

1. Primary Outcome: Physiology Measurements Before and After rTMS/Sham rTMS Protocol- Changes in Amplitude of Motor Evoked Potential (MEP) From TMS
Description: For Wrist flexion and precision grip + rTMS/Sham rTMS and Wrist extension and precision grip + rTMS/Sham rTMS we measured the changes in the MEPs before the intervention(rTMS/Sham rTMS) at minute 0, 10, 30, and 60 and then again after at minute 0, 10, 30, and 60. The information below is separated first by wrist flexion or extension, then by study visit (rTMS or Sham rTMS), and finally by subject characteristic (SCI or control). This study is a crossover design, what that means is subjects (SCI and Controls) will participate in both sessions (rTMS and Sham rTMS).
  For rTMS/Sham rTMS/Sham rTMS over control brain area we measured the changes in the MEPs at minute 0, 10, 30, and 60.The information for this arm is separated by study visit: Session 1 is rTMS, Session 2 is Sham rTMS, and Session 3 is Sham rTMS over control brain area.
  For Training + rTMS and Training + Sham rTMS we measured the changes in the MEPs at baseline, post 5 training sessions, and post all training sessions.
Time Frame: Post rTMS, Sham rTMS, and Sham rTMS over control brain for all sessions at minute 0, 10, 30, and 60
Population: The number differs due to different study visits in each arm
Measure: Mean (Standard Deviation); unit: millivolts (mV)
Groups:
- Wrist Flexion and Precision Grip + rTMS (SCI): This study arm is a crossover design. Participants will be randomized to either: Wrist flexion and precision grip + rTMS or Wrist flexion and precision grip + Sham rTMS. Participants will complete two study visits, one visit in each condition, each lasting ~2 hours separated by at least two days.
  In the Wrist flexion and precision grip + rTMS study visit, participants are asked to complete a precision grip with the index and thumb finger at the same time as flexing the wrist. Transcranial magnetic stimuli(TMS) to the brain will be administered and TMS measurements in the form of motor evoked potentials(MEPs) will be taken at minute 0, 10, 30, and 60.
  This information is from 5 SCI participants. The same 5 participants also participated in the Wrist flexion and precision grip + Sham rTMS.
- Wrist Flexion and Precision Grip + Sham rTMS (SCI): This study arm is a crossover design. Participants will be randomized to either: Wrist flexion and precision grip + rTMS or Wrist flexion and precision grip + Sham rTMS. Participants will complete two study visits, one visit in each condition, each lasting ~2 hours separated by at least two days.
  Wrist flexion and precision grip + Sham rTMS: Participants are asked to complete a precision grip with the index and thumb finger at the same time as flexing the wrist. A sham or fake magnetic stimulation to the brain (Sham rTMS) will be administered. TMS measurements in the form of motor evoked potentials (MEPs) will be taken at minute 0, 10, 30, and 60.
  This information is from 5 SCI participants. The same 5 participants also participated in the Wrist flexion and precision grip + rTMS.
- Wrist Flexion and Precision Grip + rTMS (Control): This study arm is a crossover design. Participants will be randomized to either: Wrist flexion and precision grip + rTMS or Wrist flexion and precision grip + Sham rTMS. Participants will complete two study visits, one visit in each condition, each lasting ~2 hours separated by at least two days.
  In the Wrist flexion and precision grip + rTMS study visit, participants are asked to complete a precision grip with the index and thumb finger at the same time as flexing the wrist. Transcranial magnetic stimuli(TMS) to the brain will be administered and TMS measurements in the form of motor evoked potentials(MEPs) will be taken at minute 0, 10, 30, and 60.
  This information is from 5 Control participants. The same 5 Control participants also participated in the Wrist flexion and precision grip + Sham rTMS.
- Wrist Flexion and Precision Grip + Sham rTMS (Control): This study arm is a crossover design. Participants will be randomized to either: Wrist flexion and precision grip + rTMS or Wrist flexion and precision grip + Sham rTMS. Participants will complete two study visits, one visit in each condition, each lasting ~2 hours separated by at least two days.
  Wrist flexion and precision grip + Sham rTMS: Participants are asked to complete a precision grip with the index and thumb finger at the same time as flexing the wrist. A sham or fake magnetic stimulation to the brain (Sham rTMS) will be administered. TMS measurements in the form of motor evoked potentials (MEPs) will be taken at minute 0, 10, 30, and 60.
  This information is from 5 Control participants. The same 5 Control participants also participated in the Wrist flexion and precision grip + rTMS.
- Wrist Extension and Precision Grip + rTMS (SCI): This study arm is a crossover design. Participants will be randomized to either: Wrist extension and precision grip + rTMS or Wrist extension and precision grip + Sham rTMS. Participants will complete two study visits, one visit in each condition, each lasting ~2 hours separated by at least two days.
  In the Wrist extension and precision grip + rTMS study visit, participants are asked to complete a precision grip with the index and thumb finger at the same time as extending the wrist. Transcranial magnetic stimuli(TMS) to the brain will be administered and TMS measurements in the form of motor evoked potentials(MEPs) will be taken at minute 0, 10, 30, and 60.
  This information is from 5 SCI participants. The same 5 SCI participants also participated in the Wrist extension and precision grip + Sham rTMS.
- Wrist Extension and Precision Grip + Sham rTMS (SCI): This study arm is a crossover design. Participants will be randomized to either: Wrist extension and precision grip + rTMS or Wrist extension and precision grip + Sham rTMS. Participants will complete two study visits, one visit in each condition, each lasting ~2 hours separated by at least two days.
  Wrist extension and precision grip + Sham rTMS: Participants are asked to complete a precision grip with the index and thumb finger at the same time as extending the wrist. A sham or fake magnetic stimulation to the brain (Sham rTMS) will be administered. TMS measurements in the form of motor evoked potentials (MEPs) will be taken at minute 0, 10, 30, and 60.
  This information is from 5 SCI participants. The same 5 SCI participants also participated in the Wrist extension and precision grip + rTMS.
- Wrist Extension and Precision Grip + rTMS (Control): This study arm is a crossover design. Participants will be randomized to either: Wrist extension and precision grip + rTMS or Wrist extension and precision grip + Sham rTMS. Participants will complete two study visits, one visit in each condition, each lasting ~2 hours separated by at least two days.
  In the Wrist extension and precision grip + rTMS study visit, participants are asked to complete a precision grip with the index and thumb finger at the same time as extending the wrist. Transcranial magnetic stimuli(TMS) to the brain will be administered and TMS measurements in the form of motor evoked potentials(MEPs) will be taken at minute 0, 10, 30, and 60.
  This information is from 5 Control participants. The same 5 Control participants also participated in the Wrist extension and precision grip + Sham rTMS.
- Wrist Extension and Precision Grip + Sham rTMS (Control): This study arm is a crossover design. Participants will be randomized to either: Wrist extension and precision grip + rTMS or Wrist extension and precision grip + Sham rTMS. Participants will complete two study visits, one visit in each condition, each lasting ~2 hours separated by at least two days.
  Wrist extension and precision grip + Sham rTMS: Participants are asked to complete a precision grip with the index and thumb finger at the same time as extending the wrist. A sham or fake magnetic stimulation to the brain (Sham rTMS) will be administered. TMS measurements in the form of motor evoked potentials (MEPs) will be taken at minute 0, 10, 30, and 60.
  This information is from 5 Control participants. The same 5 Control participants also participated in the Wrist extension and precision grip + rTMS.
- rTMS/Sham rTMS/Sham rTMS Over Control Brain Area: This study arm is a 3 way crossover design. Participants are randomized to one of the 3 study groups: rTMS, Sham rTMS, and Sham rTMS over control brain area. Participants will complete all study groups. Each study group consists of one study visit lasting ~2 hours and there is a 1 week washout period between each study visit.
  rTMS stimulation: In this group, rTMS stimulation will be targeting finger and wrist muscles during precision grip. TMS measurements in the form of motor evoked potentials (MEPs) will be taken at minute 0, 10, 30, and 60. The maximum voluntary contraction (MVC) will be measured using surface EMG before rTMS and again after.
  Sham or fake rTMS stimulation: In this group, Sham rTMS stimulation will be targeting finger and wrist muscles during precision grip. TMS measurements in the form of MEPs will be taken at minute 0, 10, 30, and 60. The MVC will be measured using surface EMG before rTMS and again after.
  Sham rTMS over control brain area: In this group, Sham rTMS will be applies over the dorsolateral prefrontal cortex (DLPFC) or at the leg presentation of the primary motor cortex, or at other related control area. TMS measurements in the form of MEPs will be taken at minute 0, 10, 30, and 60. The MVC will be measured using surface EMG before rTMS and again after.
  Participants are asked to wait a 1 week washout period between sessions.
  This information is from 5 SCI participants.
Arm/Group | Wrist Flexion and Precision Grip + rTMS (SCI) | Wrist Flexion and Precision Grip + Sham rTMS (SCI) | Wrist Flexion and Precision Grip + rTMS (Control) | Wrist Flexion and Precision Grip + Sham rTMS (Control) | Wrist Extension and Precision Grip + rTMS (SCI) | Wrist Extension and Precision Grip + Sham rTMS (SCI) | Wrist Extension and Precision Grip + rTMS (Control) | Wrist Extension and Precision Grip + Sham rTMS (Control) | rTMS/Sham rTMS/Sham rTMS Over Control Brain Area | Training + rTMS | Training + Sham rTMS
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 4 | 3
millivolts (mV)
  Before: minute 0: number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0 | 0
  Before: minute 0 | 0.31 (0.52) | 0.43 (0.77) | 0.45 (0.81) | 0.65 (1.12) | 0.33 (0.92) | 0.44 (0.61) | 0.59 (0.98) | 0.52 (0.83) |  |  |
  Before: minute 10: number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0 | 0
  Before: minute 10 | 0.33 (0.56) | 0.39 (0.88) | 0.47 (1.12) | 0.71 (1.08) | 0.37 (0.83) | 0.46 (0.72) | 0.66 (1.02) | 0.56 (1.06) |  |  |
  Before: minute 30: number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0 | 0
  Before: minute 30 | 0.36 (0.83) | 0.41 (0.80) | 0.51 (0.52) | 0.68 (0.91) | 0.42 (1.17) | 0.45 (0.93) | 0.63 (1.07) | 0.53 (0.92) |  |  |
  Before: minute 60: number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0 | 0
  Before: minute 60 | 0.39 (1.02) | 0.42 (0.65) | 0.53 (0.85) | 0.72 (1.15) | 0.45 (0.98) | 0.42 (1.02) | 0.65 (0.97) | 0.61 (0.82) |  |  |
  After: minute 0: number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0 | 0
  After: minute 0 | 0.36 (1.03) | 0.45 (0.81) | 0.49 (1.26) | 0.66 (0.82) | 0.44 (0.67) | 0.61 (0.98) | 0.66 (1.03) | 0.57 (0.91) |  |  |
  After: minute 10: number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0 | 0
  After: minute 10 | 0.35 (0.83) | 0.44 (0.79) | 0.51 (0.35) | 0.71 (1.13) | 0.41 (1.02) | 0.59 (1.03) | 0.71 (0.98) | 0.63 (0.70) |  |  |
  After: minute 30: number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0 | 0
  After: minute 30 | 0.50 (1.44) | 0.43 (0.61) | 0.50 (0.81) | 0.73 (0.91) | 0.42 (0.91) | 0.63 (1.12) | 0.72 (1.04) | 0.61 (1.02) |  |  |
  After: minute 60: number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0 | 0
  After: minute 60 | 0.55 (1.18) | 0.44 (0.71) | 0.55 (0.33) | 0.74 (0.78) | 0.46 (0.88) | 0.66 (0.98) | 0.74 (1.12) | 0.62 (0.87) |  |  |
  Session 1: minute 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
  Session 1: minute 0 |  |  |  |  |  |  |  |  | 0.41 (0.52) |  |
  Session 1: minute 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
  Session 1: minute 10 |  |  |  |  |  |  |  |  | 0.47 (0.91) |  |
  Session 1: minute 30: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
  Session 1: minute 30 |  |  |  |  |  |  |  |  | 0.49 (0.82) |  |
  Session 1: minute 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
  Session 1: minute 60 |  |  |  |  |  |  |  |  | 0.52 (0.70) |  |
  Session 2: minute 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
  Session 2: minute 0 |  |  |  |  |  |  |  |  | 0.59 (0.98) |  |
  Session 2: minute 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
  Session 2: minute 10 |  |  |  |  |  |  |  |  | 0.54 (0.77) |  |
  Session 2: minute 30: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
  Session 2: minute 30 |  |  |  |  |  |  |  |  | 0.61 (1.03) |  |
  Session 2: minute 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
  Session 2: minute 60 |  |  |  |  |  |  |  |  | 0.58 (0.95) |  |
  Session 3: minute 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
  Session 3: minute 0 |  |  |  |  |  |  |  |  | 0.66 (1.02) |  |
  Session 3: minute 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
  Session 3: minute 10 |  |  |  |  |  |  |  |  | 0.67 (0.98) |  |
  Session 3: minute 30: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
  Session 3: minute 30 |  |  |  |  |  |  |  |  | 0.69 (1.28) |  |
  Session 3: minute 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
  Session 3: minute 60 |  |  |  |  |  |  |  |  | 0.70 (1.02) |  |
  Baseline: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Baseline |  |  |  |  |  |  |  |  |  | 0.61 (0.79) | 0.61 (0.80)
  Post 5 training sessions: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Post 5 training sessions |  |  |  |  |  |  |  |  |  | 0.70 (0.92) | 0.68 (0.74)
  Post all training sessions: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Post all training sessions |  |  |  |  |  |  |  |  |  | 0.80 (0.83) | 0.69 (0.88)

2. Primary Outcome: Electromyography (EMG)
Description: For rTMS/Sham rTMS/Sham rTMS over control brain area we measured voluntary output in hand muscles using EMG before and after the stimulation.The information for this arm is separated by study visit: Session 1 is rTMS, Session 2 is Sham rTMS, and Session 3 is Sham rTMS over control brain area.
Time Frame: Before and After the stimulation during each 2-hour session (rTMS/Sham rTMS/Sham rTMS over control brain area)
Population: The EMG measurement was not collected in every study arm, only this arm.
Measure: Mean (Standard Deviation); unit: Millivolts (mV)
Groups:
- rTMS, Sham rTMS, Sham rTMS Over Control Brain Area: This study arm is a 3 way crossover design. Participants are randomized to one of the 3 study groups: rTMS, Sham rTMS, and Sham rTMS over control brain area. Participants will complete all study groups. Each study group consists of one study visit lasting ~2 hours and there is a 1 week washout period between each study visit.
  rTMS stimulation: In this group, rTMS stimulation will be targeting finger and wrist muscles during precision grip. TMS measurements in the form of motor evoked potentials (MEPs) will be taken at minute 0, 10, 30, and 60. The maximum voluntary contraction (MVC) will be measured using surface EMG before rTMS and again after.
  Sham or fake rTMS stimulation: In this group, Sham rTMS stimulation will be targeting finger and wrist muscles during precision grip. TMS measurements in the form of MEPs will be taken at minute 0, 10, 30, and 60. The MVC will be measured using surface EMG before rTMS and again after.
  Sham rTMS over control brain area: In this group, Sham rTMS will be applies over the dorsolateral prefrontal cortex (DLPFC) or at the leg presentation of the primary motor cortex, or at other related control area. TMS measurements in the form of MEPs will be taken at minute 0, 10, 30, and 60. The MVC will be measured using surface EMG before rTMS and again after.
  Participants are asked to wait a 1 week washout period between sessions.
  This information is from 5 SCI participants.
Arm/Group | rTMS, Sham rTMS, Sham rTMS Over Control Brain Area
Number analyzed (Participants) | 5
Millivolts (mV)
  Session 1: Before | 0.138 (0.239)
  Session 1: After | 0.191 (0.323)
  Session 2: Before | 0.204 (0.361)
  Session 2: After | 0.208 (0.384)
  Session 3: Before | 0.221 (0.329)
  Session 3: After | 0.231 (0.352)

3. Secondary Outcome: The Jebsen Taylor Hand Function Test (JTT)
Description: The JTT is a standardized test of several major aspects of hand function using simulated activities of daily living (writing, picking up small objects, picking up heavy objects etc.). The time taken to perform simulated activities of daily living is assessed. Lesser time to perform the activities would be considered a better outcome.
Time Frame: The JTT was measured at Baseline, Post 5 training sessions, and Post all training sessions at each 2-hour session.
Population: The JTT was not measured in all study arms, only this arm.
Measure: Mean (Standard Deviation); unit: Time (seconds)
Groups:
- Training + rTMS: Participants are asked to follow a target line on the computer as accurately as possible while performing precision grips. Magnetic stimulation will be given during. Participants are asked to complete 10 of these sessions. Participants will also be asked to complete measurements at Baseline, Post 5 training sessions, and Post all training sessions.
- Training + Sham rTMS: Participants are asked to follow a target line on the computer as accurately as possible while performing precision grips. Sham or fake Magnetic stimulation will be given during. Participants are asked to complete 10 of these sessions. Participants will also be asked to complete measurements at Baseline, Post 5 training sessions, and Post all training sessions.
Arm/Group | Training + rTMS | Training + Sham rTMS
Number analyzed (Participants) | 4 | 3
Time (seconds)
  Baseline | 74.1 (21.6) | 88.6 (19.6)
  Post 5 training sessions | 54.4 (13.9) | 79.3 (18.7)
  Post all training sessions | 44.8 (15.2) | 84.8 (14.2)

ADVERSE EVENTS:
Time Frame: The adverse event data was collected from baseline to completion of study visits for each participant, an average of 6 days for Arm 1 and an average of 3 weeks for Arm 2 and 3.
Groups:
- Training + rTMS: Participants will be asked to follow a target line on the computer as accurately as possible while performing precision grips or foot movement. Magnetic stimulation will be given during rest and movement.
  rTMS: small magnetic pulses will be given to the brain in a non invasive manner.
  Training: at the direction of the researcher the participant will be instructed to do repetitive motor movements with their arm, hand or leg. This is called training
- Training + Sham rTMS: Participants will be asked to follow a target line on the computer as accurately as possible while performing precision grips or foot movement. Magnetic stimulation will be given during rest and movement.
  Sham rTMS: sham or fake stimulation (TMS or rTMS) will be given to the brain in a non invasive manner
  Training: at the direction of the researcher the participant will be instructed to do repetitive motor movements with their arm, hand or leg. This is called training
Arm/Group | Wrist Flexion and Precision Grip + rTMS and Sham rTMS | Wrist Extension and Precision Grip + rTMS and Sham rTMS | rTMS/Sham rTMS/Sham rTMS Over Control Brain Area | Training + rTMS | Training + Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/5 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/5 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/5 | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT01915095/Prot_SAP_000.pdf